CLINICAL TRIAL: NCT04102540
Title: Information Visualizations to Facilitate HIV-related Patient-provider Communication in New York City (Info Viz: HIV-NYC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Associate Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAS4611; 1K99NR017829-01A1 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Health Communication
Keywords: Information Visualization

STUDY DESIGN:
Intervention Model Description: This study will use a single pretest-posttest design to evaluate if using infographics for patient education can lead to improved patient outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infographic intervention group (Experimental): Participants in the infographic intervention group will receive health education using infographics during a study visit scheduled immediately following their regularly scheduled clinic visits.
  Interventions: Other: Infographic intervention

INTERVENTIONS:
Other: Infographic intervention — Information visualizations (infographics) will be used to teach participants about HIV during study visits immediately following their normal clinic visits.

SUMMARY:
To complete the study aims, a mixed methods study that includes a single group pretest-posttest study design will be used to pilot test the infographic intervention. In-depth interviews will be completed with a selection of participants to explore participant perceptions of HIV-related communication using infographics. Data will be collected from participants through baseline (at enrollment) and follow up assessments at 3- and 6-month follow up visits). Follow up interviews will be conducted with members of the clinical team to ascertain their perspectives on the clinical utility of infographics.

DETAILED DESCRIPTION:
Latinos are the largest and fastest growing minority group in the US, and they are disproportionately affected by HIV. In 2014, almost 25% of new cases of HIV infections were among Latinos although they only represent 17% of the US population. Additionally, Latinos have a faster rate of progression from HIV to AIDS, higher rates of HIV-related deaths, and marked delay in the diagnosis of infections. Approximately 42% of HIV diagnoses among Latinos in the US are in persons born abroad. In absolute numbers, new HIV diagnoses among foreign-born individuals in the US were the highest among Caribbean-born persons, which may partially be attributed to high rates of bidirectional travel. It is, therefore, critical that HIV prevention and treatment activities incorporate factors associated with Latino immigrant and transnational groups. In Washington Heights, New York City, understanding these factors related with bi-directional travel to the Dominican Republic (DR) is warranted, as the Latino population of Washington Heights is largely comprised of Dominicans.

Many factors contribute to the health disparities experienced by Latinos, of which low health literacy and literacy in general are potential contributors. Health literacy, or "the degree to which individuals have the capacity to obtain, process, and understand basic health information and services needed to make appropriate health decisions," is an established concern affecting vulnerable communities globally. Not surprisingly, Spanish-speaking, less educated, and/or foreign-born Latinos have lower health literacy than those born in the US. Low health literacy can lead to worse health outcomes, less use of services, and poorer knowledge of illness. Also, patients with limited health literacy are likely to have low numeracy which affects interpretations of medication quantities, time between doses, and time between appointments, among other quantitative knowledge relating to effective management of HIV.

Infographics are emerging technologies to help teach complex health concepts to patients with low health literacy. When effectively designed, infographics (information visualizations) contain a depth and breadth of information and lead to improved understanding of concepts. By carefully selecting the design and included content, simple images can convey large amounts of information in a visually appealing and comprehensible way. Methodically constructed infographics have been shown to improve communication about health behaviors and health risks and minimize comprehension differences between individuals with high and low health literacy. They can also help improve information exchange amidst culture and language differences by using images familiar to patients to explain complicated processes as well as augment attention span and recall of learned material. Furthermore, rigorously designed and evaluated infographics can help mitigate health disparities by helping clinicians provide the information that people need for effective health management in an understandable way.

During preliminary studies, the investigators developed a set of infographics designed to facilitate HIV-related clinician-patient communication during clinic visits. Initial infographics were designed by persons living with HIV (PLWH) in the Dominican Republic and are now being tested for feasibility and usability among a cohort in the DR. In this study, the investigators propose to assess the feasibility of using the infographic intervention in a clinic that specializes in HIV care in Washington Heights to improve clinical communication and subsequently, patient outcomes. Additionally, the investigators will collect information about acculturation and bi-directional travel to more thoroughly assess how these factors relate to HIV infection among Hispanic/Latino populations living in the US.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age
* Living with HIV and has a detectable viral load
* Self-identifies as Hispanic/Latino
* Plan to receive care at the same clinic for the next 6 months

Exclusion Criteria:

* Does not meet inclusion criteria
* Not able to understand study procedures or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, RN, Principal Investigator — Columbia University; Samantha B Stonbraker, PhD, MPH, RN, Study Director — Columbia University
Locations (1):
- Comprehensive HIV Program of NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participant data will be made available to qualified researchers seeking to replicate methods or to those working on a new study who need the evidence-base to do so in a rigorous way. All de-identified participant data will be shared with other researchers. Please note that much of this data will be in Spanish.
Supporting Information: CSR, Analytic Code
Time Frame: Data will be available 3 months after the publication of primary results.
Access Criteria: To request data please email the study director listed on this record with the reason you need the data and your planned use of it.

REFERENCES:
- [Background] Passel J, Cohn D, Lopez M. Hispanics account for more than half of nation's growth in past decade. Washington DC: Pew Hispanic Center;2011.
- [Background] Brown A, Hugo Lopez M. Mapping the Latino Population, By State, County and City. Washington DC2013.
- [Background] Henao-Martinez AF, Castillo-Mancilla JR. The Hispanic HIV Epidemic. Curr Infect Dis Rep. 2013 Feb;15(1):46-51. doi: 10.1007/s11908-012-0306-0. PMID 23184612
- [Background] Gonzalez JS, Hendriksen ES, Collins EM, Duran RE, Safren SA. Latinos and HIV/AIDS: examining factors related to disparity and identifying opportunities for psychosocial intervention research. AIDS Behav. 2009 Jun;13(3):582-602. doi: 10.1007/s10461-008-9402-4. Epub 2008 May 23. PMID 18498050
- [Background] Xia Q, Braunstein SL, Wiewel EW, Hadler JL, Torian LV. Persistent Racial Disparities in HIV Infection in the USA: HIV Prevalence Matters. J Racial Ethn Health Disparities. 2017 Feb;4(1):87-93. doi: 10.1007/s40615-015-0205-9. Epub 2016 Jan 8. PMID 26746424
- [Background] Lescano CM, Brown LK, Raffaelli M, Lima LA. Cultural factors and family-based HIV prevention intervention for Latino youth. J Pediatr Psychol. 2009 Nov-Dec;34(10):1041-52. doi: 10.1093/jpepsy/jsn146. Epub 2009 Jan 30. PMID 19181820
- [Background] Centers for Disease Control and Prevention. HIV in the United States: At a Glance. 2015; https://www.cdc.gov/hiv/statistics/overview/ataglance.html. Accessed June, 2017.
- [Background] Vega WA, Rodriguez MA, Gruskin E. Health disparities in the Latino population. Epidemiol Rev. 2009;31:99-112. doi: 10.1093/epirev/mxp008. Epub 2009 Aug 27. PMID 19713270
- [Background] Prosser AT, Tang T, Hall HI. HIV in persons born outside the United States, 2007-2010. JAMA. 2012 Aug 8;308(6):601-7. doi: 10.1001/jama.2012.9046. PMID 22820630
- [Background] Wiewel EW, Torian LV, Hanna DB, Bocour A, Shepard CW. Foreign-Born Persons Diagnosed with HIV: Where are They From and Where Were They Infected? AIDS Behav. 2015 May;19(5):890-8. doi: 10.1007/s10461-014-0954-1. PMID 25524308
- [Background] Gill MJ, Krentz HB. Unappreciated epidemiology: the churn effect in a regional HIV care programme. Int J STD AIDS. 2009 Aug;20(8):540-4. doi: 10.1258/ijsa.2008.008422. PMID 19625584
- [Background] Saint-Jean G, Devieux J, Malow R, Tammara H, Carney K. Substance Abuse, Acculturation, and HIV Risk among Caribbean-Born Immigrants in the United States. J Int Assoc Physicians AIDS Care (Chic). 2011 Sep-Oct;10(5):326-32. doi: 10.1177/1545109711401749. Epub 2011 Apr 21. PMID 21511982
- [Background] McMahon T, Ward PR. HIV among immigrants living in high-income countries: a realist review of evidence to guide targeted approaches to behavioural HIV prevention. Syst Rev. 2012 Nov 20;1:56. doi: 10.1186/2046-4053-1-56. PMID 23168134
- [Background] Shedlin MG, Drucker E, Decena CU, Hoffman S, Bhattacharya G, Beckford S, Barreras R. Immigration and HIV/AIDS in the New York Metropolitan Area. J Urban Health. 2006 Jan;83(1):43-58. doi: 10.1007/s11524-005-9006-5. PMID 16736354
- [Background] Nwosu C, Balaova J. Immigrants from the Dominican Republic in the United States. 2014; https://www.migrationpolicy.org/article/immigrants-dominican-republic-united-states. Accessed May, 2019.
- [Background] Osborn CY, Paasche-Orlow MK, Davis TC, Wolf MS. Health literacy: an overlooked factor in understanding HIV health disparities. Am J Prev Med. 2007 Nov;33(5):374-8. doi: 10.1016/j.amepre.2007.07.022. PMID 17950402
- [Background] Wawrzyniak AJ, Ownby RL, McCoy K, Waldrop-Valverde D. Health literacy: impact on the health of HIV-infected individuals. Curr HIV/AIDS Rep. 2013 Dec;10(4):295-304. doi: 10.1007/s11904-013-0178-4. PMID 24222474
- [Background] Laws MB, Lee Y, Rogers WH, Beach MC, Saha S, Korthuis PT, Sharp V, Cohn J, Moore R, Wilson IB. Provider-patient communication about adherence to anti-retroviral regimens differs by patient race and ethnicity. AIDS Behav. 2014 Jul;18(7):1279-87. doi: 10.1007/s10461-014-0697-z. PMID 24464408
- [Background] Sentell TL, Halpin HA. Importance of adult literacy in understanding health disparities. J Gen Intern Med. 2006 Aug;21(8):862-6. doi: 10.1111/j.1525-1497.2006.00538.x. PMID 16881948
- [Background] Koskan A, Friedman D, Messias D. Health literacy among Hispanics: a systematic research review (1992-2008). Hispanic Health Care International. 2010;8:65-76.
- [Background] Paasche-Orlow MK, Parker RM, Gazmararian JA, Nielsen-Bohlman LT, Rudd RR. The prevalence of limited health literacy. J Gen Intern Med. 2005 Feb;20(2):175-84. doi: 10.1111/j.1525-1497.2005.40245.x. PMID 15836552
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Kalichman SC, Rompa D. Functional health literacy is associated with health status and health-related knowledge in people living with HIV-AIDS. J Acquir Immune Defic Syndr. 2000 Dec 1;25(4):337-44. doi: 10.1097/00042560-200012010-00007. PMID 11114834
- [Background] Garcia-Retamero R, Galesic M. Communicating treatment risk reduction to people with low numeracy skills: a cross-cultural comparison. Am J Public Health. 2009 Dec;99(12):2196-202. doi: 10.2105/AJPH.2009.160234. Epub 2009 Oct 15. PMID 19833983
- [Background] Moore JO, Boyer EW, Safren S, Robbins GK, Boudreaux ED, Rosen R, Barton B, Moss F. Designing interventions to overcome poor numeracy and improve medication adherence in chronic illness, including HIV/AIDS. J Med Toxicol. 2011 Jun;7(2):133-8. doi: 10.1007/s13181-011-0149-3. PMID 21455810
- [Background] Dowse R, Ramela T, Browne SH. An illustrated leaflet containing antiretroviral information targeted for low-literate readers: development and evaluation. Patient Educ Couns. 2011 Dec;85(3):508-15. doi: 10.1016/j.pec.2011.01.013. Epub 2011 Feb 8. PMID 21306856
- [Background] Garcia-Retamero R, Okan Y, Cokely ET. Using visual aids to improve communication of risks about health: a review. ScientificWorldJournal. 2012;2012:562637. doi: 10.1100/2012/562637. Epub 2012 May 2. PMID 22629146
- [Background] McCaffery KJ, Dixon A, Hayen A, Jansen J, Smith S, Simpson JM. The influence of graphic display format on the interpretations of quantitative risk information among adults with lower education and literacy: a randomized experimental study. Med Decis Making. 2012 Jul-Aug;32(4):532-44. doi: 10.1177/0272989X11424926. Epub 2011 Nov 10. PMID 22074912
- [Background] Ancker JS, Senathirajah Y, Kukafka R, Starren JB. Design features of graphs in health risk communication: a systematic review. J Am Med Inform Assoc. 2006 Nov-Dec;13(6):608-18. doi: 10.1197/jamia.M2115. Epub 2006 Aug 23. PMID 16929039
- [Background] Arcia A, Suero-Tejeda N, Bales ME, Merrill JA, Yoon S, Woollen J, Bakken S. Sometimes more is more: iterative participatory design of infographics for engagement of community members with varying levels of health literacy. J Am Med Inform Assoc. 2016 Jan;23(1):174-83. doi: 10.1093/jamia/ocv079. Epub 2015 Jul 13. PMID 26174865
- [Background] Houts PS, Doak CC, Doak LG, Loscalzo MJ. The role of pictures in improving health communication: a review of research on attention, comprehension, recall, and adherence. Patient Educ Couns. 2006 May;61(2):173-90. doi: 10.1016/j.pec.2005.05.004. Epub 2005 Aug 24. PMID 16122896
- [Background] Kasper J, van de Roemer A, Pottgen J, Rahn A, Backhus I, Bay Y, Kopke S, Heesen C. A new graphical format to communicate treatment effects to patients-A web-based randomized controlled trial. Health Expect. 2017 Aug;20(4):797-804. doi: 10.1111/hex.12522. Epub 2016 Dec 16. PMID 27981688
- [Background] Garcia-Retamero R, Dhami MK. Pictures speak louder than numbers: on communicating medical risks to immigrants with limited non-native language proficiency. Health Expect. 2011 Mar;14 Suppl 1(Suppl 1):46-57. doi: 10.1111/j.1369-7625.2011.00670.x. PMID 21323820
- [Background] Katz MG, Jacobson TA, Veledar E, Kripalani S. Patient literacy and question-asking behavior during the medical encounter: a mixed-methods analysis. J Gen Intern Med. 2007 Jun;22(6):782-6. doi: 10.1007/s11606-007-0184-6. Epub 2007 Apr 12. PMID 17431697
- [Background] Zikmund-Fisher BJ, Witteman HO, Dickson M, Fuhrel-Forbis A, Kahn VC, Exe NL, Valerio M, Holtzman LG, Scherer LD, Fagerlin A. Blocks, ovals, or people? Icon type affects risk perceptions and recall of pictographs. Med Decis Making. 2014 May;34(4):443-53. doi: 10.1177/0272989X13511706. Epub 2013 Nov 18. PMID 24246564
- [Background] Cuellar I, Arnold B, Maldonado RJHjobs. Acculturation rating scale for Mexican Americans-II: A revision of the original ARSMA scale. 1995;17(3):275-304.
- [Background] Cuellar I, Bastida E, Braccio SM. Residency in the United States, subjective well-being, and depression in an older Mexican-origin sample. J Aging Health. 2004;16(4):447-66. doi: 10.1177/0898264304265764. PMID 15271265
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Kallio H, Pietila AM, Johnson M, Kangasniemi M. Systematic methodological review: developing a framework for a qualitative semi-structured interview guide. J Adv Nurs. 2016 Dec;72(12):2954-2965. doi: 10.1111/jan.13031. Epub 2016 Jun 23. PMID 27221824
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] McSweeney JC, Allan JD, Mayo K. Exploring the use of explanatory models in nursing research and practice. Image J Nurs Sch. 1997;29(3):243-8. doi: 10.1111/j.1547-5069.1997.tb00992.x. PMID 9378479
- [Background] Sandelowski M. Sample size in qualitative research. Res Nurs Health. 1995 Apr;18(2):179-83. doi: 10.1002/nur.4770180211. PMID 7899572
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] White MD, Marsh EE. Content analysis: A flexible methodology. Library trends. 2006;55(1):22-45.
- [Background] Kleinman A, Eisenberg L, Good B. Culture, illness, and care: clinical lessons from anthropologic and cross-cultural research. Ann Intern Med. 1978 Feb;88(2):251-8. doi: 10.7326/0003-4819-88-2-251. PMID 626456
- [Background] Gioia DA, Corley KG, Hamilton AL. Seeking qualitative rigor in inductive research: Notes on the Gioia methodology. Organizational research methods. 2013;16(1):15-31.
- [Background] Berkhof M, van Rijssen HJ, Schellart AJ, Anema JR, van der Beek AJ. Effective training strategies for teaching communication skills to physicians: an overview of systematic reviews. Patient Educ Couns. 2011 Aug;84(2):152-62. doi: 10.1016/j.pec.2010.06.010. Epub 2010 Jul 29. PMID 20673620
- [Background] Dickens A, Utley-Smith Q, Stott G, Relf M. Evaluation of communication techniques used by HIV specialty providers caring for patients with low health literary in an outpatient HIV clinical setting. Journal of Nursing Education & Practice. 2013;3(7)
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] Toren KG, Buskin SE, Dombrowski JC, Cassels SL, Golden MR. Time From HIV Diagnosis to Viral Load Suppression: 2007-2013. Sex Transm Dis. 2016 Jan;43(1):34-40. doi: 10.1097/OLQ.0000000000000376. PMID 26650994
- [Background] Nash D, Katyal M, Brinkhof MW, Keiser O, May M, Hughes R, Dabis F, Wood R, Sprinz E, Schechter M, Egger M; ART-LINC Collaboration of IeDEA. Long-term immunologic response to antiretroviral therapy in low-income countries: a collaborative analysis of prospective studies. AIDS. 2008 Nov 12;22(17):2291-302. doi: 10.1097/QAD.0b013e3283121ca9. PMID 18981768
- [Background] Street RL Jr, Makoul G, Arora NK, Epstein RM. How does communication heal? Pathways linking clinician-patient communication to health outcomes. Patient Educ Couns. 2009 Mar;74(3):295-301. doi: 10.1016/j.pec.2008.11.015. Epub 2009 Jan 15. PMID 19150199
- [Background] Glanz K, Rimer BK, Viswanath K. Health behavior and health education: theory, research, and practice. Fourth ed: John Wiley & Sons; 2008.
- [Background] Dang BN, Westbrook RA, Hartman CM, Giordano TP. Retaining HIV Patients in Care: The Role of Initial Patient Care Experiences. AIDS Behav. 2016 Oct;20(10):2477-2487. doi: 10.1007/s10461-016-1340-y. PMID 26910339
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; GEEMA Study Group. Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. AIDS. 2002 Mar 8;16(4):605-13. doi: 10.1097/00002030-200203080-00012. PMID 11873004
- [Background] Schnall R, Liu J, Cho H, Hirshfield S, Siegel K, Olender S. A Health-Related Quality-of-Life Measure for Use in Patients with HIV: A Validation Study. AIDS Patient Care STDS. 2017 Feb;31(2):43-48. doi: 10.1089/apc.2016.0252. Epub 2017 Jan 4. PMID 28051875
- [Background] Lee SY, Stucky BD, Lee JY, Rozier RG, Bender DE. Short Assessment of Health Literacy-Spanish and English: a comparable test of health literacy for Spanish and English speakers. Health Serv Res. 2010 Aug;45(4):1105-20. doi: 10.1111/j.1475-6773.2010.01119.x. Epub 2010 May 24. PMID 20500222
- [Background] McGuire WJ. McGuire's classic input-output framework for constructing persuasive messages. Public communication campaigns. 2013;4:133-145.
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Osborn CY, Weiss BD, Davis TC, Skripkauskas S, Rodrigue C, Bass PF, Wolf MS. Measuring adult literacy in health care: performance of the newest vital sign. Am J Health Behav. 2007 Sep-Oct;31 Suppl 1:S36-46. doi: 10.5555/ajhb.2007.31.supp.S36. PMID 17931135

RESULTS

PARTICIPANT FLOW:
Groups:
- Infographic Intervention Group: Participants in the intervention group will receive health education using infographics (Infographic Intervention) during a study visit scheduled immediately following their regularly scheduled clinic visits.
  Infographic intervention: Information visualizations (infographics) will be used to teach participants about HIV during study visits immediately following their normal clinic visits.
Period: Overall Study
Arm/Group | Infographic Intervention Group
Started | 32
Completed | 24
Not Completed | 8
Not completed — Withdrawn by PI | 2
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Two participants were removed from the study by the PI. Their information was not included in the calculations of participants' characteristics at baseline.
Groups:
- Intervention Group: Participants in the intervention group will receive health education using infographics (Infographic Intervention) during a study visit scheduled immediately following their regularly scheduled clinic visits.
  Infographic intervention: Information visualizations (infographics) will be used to teach participants about HIV during study visits immediately following their normal clinic visits.
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (14.19)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 18
  Female | 11
  Other | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 12
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Country of birth [Count of Participants; unit: Participants]
  United States | 9
  Dominican Republic | 15
  Other | 6
Married or in a serious relationship [Count of Participants; unit: Participants]
  Married or in a serious relationship | 7
  NOT married or in a serious relationship | 23
Highest level of education completed [Count of Participants; unit: Participants]
  0-5 years of school | 4
  6-8 years of school | 6
  9-11 years of school | 6
  Finished HS/ has GED | 10
  University or other education past HS | 4
New Patient [Count of Participants; unit: Participants]
  New patient | 4
  Established patient | 26
Years living with HIV [Mean (Standard Deviation); unit: Years] | 16.28 (9.7)
Years attending the clinic [Mean (Standard Deviation); unit: Years] | 10.04 (9.41)
Preferred language of participation [Count of Participants; unit: Participants]
  English-speaking | 12
  Spanish-speaking | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean CD4 Count
Description: Mean Cluster of Differentiation 4 (CD4) count at each time point.
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn by the PI and were not included in analyses.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Cells/mm^3
  CD4 Count at Baseline | 321.5 (1038)
  CD4 Count after second exposure to intervention: number analyzed (Participants) | 27
  CD4 Count after second exposure to intervention | 418 (944)
  CD4 Count after third exposure to intervention: number analyzed (Participants) | 19
  CD4 Count after third exposure to intervention | 390.5 (834)
Statistical Analysis 1: Comparison: Infographic Intervention Group; Statistical analysis of CD4 count between baseline/exposure 1 and exposure 2 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median CD4 count at baseline/exposure 1 was exactly equivalent to the median CD4 count following exposure 2 to the intervention; p = 0.283, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 57.39, 95% CI 2-sided [-48.9 to 163.7] — This is the difference in median CD4 count between baseline/exposure 1 and exposure 2
Statistical Analysis 2: Comparison: Infographic Intervention Group; Statistical analysis of CD4 count between baseline/exposure 1 and exposure 3 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median CD4 count at baseline/exposure 1 was exactly equivalent to the median CD4 count following the exposure 3 to the intervention; p = 0.1823, Quantile regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 60.83, 95% CI 2-sided [-29.5 to 151.2] — This is the difference in median CD4 count between baseline/exposure 1 and exposure 3

2. Primary Outcome: Mean Viral Load
Description: Mean viral load at each time point
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
copies/mL
  Baseline/exposure 1 | 97,266 (340,644)
  Exposure 2: number analyzed (Participants) | 27
  Exposure 2 | 93,242 (286,207)
  Exposure 3: number analyzed (Participants) | 19
  Exposure 3 | 21,116 (79,176)
Statistical Analysis 1: Comparison: Infographic Intervention Group; Statistical analysis of viral load between baseline/exposure 1 and exposure 2 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median viral load at baseline/exposure 1 was exactly equivalent to the median viral load following exposure 2 to the intervention; p = 0.7795, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Median Difference (Net) = -42, 95% CI 2-sided [-339.8 to 255.8] — This is the difference in median viral load between baseline/exposure 1 and exposure 2
Statistical Analysis 2: Comparison: Infographic Intervention Group; Statistical analysis of viral load between baseline/exposure 1 and exposure 3 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median viral load at baseline/exposure 1 was exactly equivalent to the median viral load following exposure 3 to the intervention; p = 0.5971, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Median Difference (Net) = -63.00, 95% CI 2-sided [-296.1 to 170.1]; This is the difference in median viral load between baseline/exposure 1 and exposure 3

3. Secondary Outcome: Mean Score on HIV-related Knowledge Assessment
Description: 14 questions pertaining to HIV-related knowledge were developed according to the information that will be included in the intervention. Participants will receive one point for each correct answer and then the scores for each question will be summed to obtain a final score. Therefore, the minimum score will be 0 and maximum score will be 14 where the scores closer to 14 indicate patients have more HIV-related knowledge.
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
score on a scale
  Baseline/exposure 1 | 10.10 (2.43)
  Exposure 2: number analyzed (Participants) | 27
  Exposure 2 | 12.23 (1.51)
  Exposure 3: number analyzed (Participants) | 19
  Exposure 3 | 12.21 (1.59)
Statistical Analysis 1: Comparison: Infographic Intervention Group; Statistical analysis of HIV-related knowledge scores between baseline/exposure 1 and exposure 2 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median HIV-related knowledge score at baseline/exposure 1 was exactly equivalent to the median HIV-related knowledge score following exposure 2 to the intervention; p < .0001, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 2.12, 95% CI 2-sided [1.2 to 3.0] — This is the difference in median HIV-Related knowledge scores between baseline/exposure 1 and exposure 2
Statistical Analysis 2: Comparison: Infographic Intervention Group; Statistical analysis of HIV-related knowledge scores between baseline/exposure 1 and exposure 3 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median HIV-related knowledge score at baseline/exposure 1 was exactly equivalent to the median HIV-related knowledge score following exposure 3 to the intervention; p < .0001, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 2.00, 95% CI 2-sided [1.2 to 2.8] — This is the difference in median HIV-related knowledge score between baseline/exposure 1 and exposure 3

4. Secondary Outcome: Mean Score on Satisfaction With Care Scale
Description: 7 questions on patients' satisfaction with health care provider and the health care center adapted from previously validated instruments were included.
  Each question response from included questions has a different score range:
  Question 1: 1 - 7 Question 2: 1 - 10 Question 3: 1 - 7 Question 4: 1 - 5 Question 5: 1 - 7 Question 6: 1 - 7 Question 7: 1 - 5
  Total scores range from 7 - 48, which is calculated from the lowest and highest possible scores on each of the included questions. Higher scores indicating more satisfaction with care.
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
score on a scale
  Baseline/exposure 1 | 44.93 (3.40)
  Exposure 2: number analyzed (Participants) | 27
  Exposure 2 | 45.18 (2.81)
  Exposure 3: number analyzed (Participants) | 19
  Exposure 3 | 44.29 (5.06)

5. Secondary Outcome: Mean Score on the SEMCD Scale
Description: The Self-Efficacy for Managing Chronic Disease (SEMCD) scale is a 6-item questionnaire that measures confidence in one's ability to manage fatigue, pain, emotional distress, and other symptoms using self-management techniques. Each item is scored from a minimum value of 1 which indicates "not at all confident" to a maximum score of 10, which indicates "completely confident." Final scores are calculated as the mean of the 6 questions ranging from 1(minimum) to 10 (maximum), where higher scores indicate higher self-efficacy (better outcome).
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
score on a scale
  Baseline/exposure 1 | 8.01 (1.72)
  Exposure 2: number analyzed (Participants) | 27
  Exposure 2 | 8.13 (1.46)
  Exposure 3: number analyzed (Participants) | 19
  Exposure 3 | 8.48 (1.89)
Statistical Analysis 1: Comparison: Infographic Intervention Group; Statistical analysis of self-efficacy to manage HIV scale score between baseline/exposure 1 and exposure 2 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median self-efficacy to manage HIV scale score at baseline/exposure 1 was exactly equivalent to the median self-efficacy to manage HIV scale score following exposure 2 to the intervention; p = 0.9879, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 0.01, 95% CI 2-sided [-0.7 to 0.7] — This is the difference in median self-efficacy to manage HIV scale scores between baseline/exposure 1 and exposure 2
Statistical Analysis 2: Comparison: Infographic Intervention Group; Statistical analysis of self-efficacy to manage HIV scale score between baseline/exposure 1 and exposure 3 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median self-efficacy to manage HIV scale score at baseline/exposure 1 was exactly equivalent to the median self-efficacy to manage HIV scale score following exposure 3 to the intervention; p = 0.1550, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 0.57, 95% CI 2-sided [-0.2 to 1.4] — This is the difference in median self-efficacy to manage HIV scale scores between baseline/exposure 1 and exposure 3

6. Secondary Outcome: Number of Participants Who Are Adherent to Their Medications
Description: Adherence will be measured with the validated simplified medication adherence questionnaire (SMAQ)-6 scale, a 6-item questionnaire. A person is considered "non-adherent" if there is a "yes" answer for any of items 1,2,3, and 5. Additionally, if they answer that they have missed more than two doses of their medication in the past week (item 4) or if they have gone more than two days without taking their medication in the past 3 months (item 6), they are also considered "non-adherent."
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Participants
  Baseline/exposure 1: Adherent | 10
  Baseline/exposure 1: Non-adherent | 20
  Baseline/exposure 1: Missing | 0
  Exposure 2: Adherent | 7
  Exposure 2: Non-adherent | 15
  Exposure 2: Missing | 8
  Exposure 3: Adherent | 11
  Exposure 3: Non-adherent | 13
  Exposure 3: Missing | 6
Statistical Analysis 1: Comparison: Infographic Intervention Group; For analysis, we dichotomized participants adherence as "adherent" or "non-adherent."; Test type: Other — In this model, the null hypothesis was that the odds of being non-adherent at baseline/exposure 1 were exactly equal to the odds of being non-adherent at exposure 2 giving an odds ratio of one for the null hypothesis; p = 0.8190, Regression, Logistic — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; This model included random effects for subjects; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.30 to 4.52] — In this model, the odds ratio estimate is for the odds of being non-adherent at exposure 2 relative to the odds of being non-adherent at baseline/exposure 1
Statistical Analysis 2: Comparison: Infographic Intervention Group; For analysis, we dichotomized participants adherence as "adherent" or "non-adherent."; Test type: Other — In this model, the null hypothesis was that the odds of being non-adherent at baseline/exposure 1 were exactly equal to the odds of being non-adherent at exposure 3 giving an odds ratio of one for the null hypothesis; p = 0.1332, Regression, Logistic — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; This model included random effects for subjects; Odds Ratio (OR) = 0.3, 95% CI 2-sided [0.07 to 1.43] — In this model, the odds ratio estimate is for the odds of being non-adherent at exposure 3 relative to the odds of being non-adherent at baseline/exposure 1

7. Secondary Outcome: Number of Participants Who Reported Each of the 5 General Health Categories
Description: Participants rated their general health as "excellent," "very good," "good," "more or less," or "bad."
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Participants
  Baseline/exposure 1: Bad | 1
  Baseline/exposure 1: More or less | 15
  Baseline/exposure 1: Good | 6
  Baseline/exposure 1: Very Good | 4
  Baseline/exposure 1: Excellent | 4
  Baseline/exposure 1: Missing | 0
  Exposure 2: Bad | 0
  Exposure 2: More or less | 10
  Exposure 2: Good | 7
  Exposure 2: Very Good | 1
  Exposure 2: Excellent | 4
  Exposure 2: Missing | 8
  Exposure 3: Bad | 0
  Exposure 3: More or less | 11
  Exposure 3: Good | 5
  Exposure 3: Very Good | 4
  Exposure 3: Excellent | 4
  Exposure 3: Missing | 6
Statistical Analysis 1: Comparison: Infographic Intervention Group; For analysis, we dichotomized participants' responses into the following categories: "good" vs "bad" health, where "good" included participant responses: "excellent," "very good," "good," and "bad" included the participant responses: "more or less" and "bad."; Test type: Other — In this model, the null hypothesis was that the odds of good health at baseline/exposure 1 were exactly equal to the odds of good health at exposure 2 giving an odds ratio of one for the null hypothesis; p = 0.3160, Regression, Logistic — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; This model included random effects for subjects; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.57 to 5.46] — This is the estimated odds ratio of having good health at exposure 2 relative to baseline/exposure 1
Statistical Analysis 2: Comparison: Infographic Intervention Group; [analysis description as in outcome 7, analysis 1]; Test type: Other — In this model, the null hypothesis was that the odds of having good health at baseline/exposure 1 were exactly equal to the odds of having good health at exposure 3 giving an odds ratio of one for the null hypothesis; p = 0.8609, Regression, Logistic — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; This model included random effects for subjects; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.32 to 3.93] — This is the estimated odds ratio of having good health at exposure 3 relative to baseline/exposure 1

8. Secondary Outcome: Mean Score on Current Health Status
Description: Current health status will be assessed with one question from the Health Status Assessment which asks participants to rate their current health by providing a number on a scale from 0 - 100 where 0=death or worst possible health and 100=perfect or best possible health.
Time Frame: Baseline, 3-, and 6-months
Population: 2 participants were withdrawn from the study by the PI, therefore, 30 subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
score on a scale
  Baseline/exposure 1 | 68 (20.66)
  Exposure 2: number analyzed (Participants) | 27
  Exposure 2 | 75.45 (17.03)
  Exposure 3: number analyzed (Participants) | 19
  Exposure 3 | 82.29 (16.8)
Statistical Analysis 1: Comparison: Infographic Intervention Group; Statistical analysis of current health status between baseline/exposure 1 and exposure 2 to the intervention; Test type: Other — In this analysis, our null hypothesis was that the median current health status at baseline/exposure 1 was exactly equivalent to the median current health status following exposure 2 to the intervention; p = 0.0572, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 9.13, 95% CI 2-sided [-0.3 to 18.6] — This is the difference in median current health status between baseline/exposure 1 and exposure 2
Statistical Analysis 2: Comparison: Infographic Intervention Group; [analysis description as in outcome 5, analysis 2]; Test type: Other — In this analysis, our null hypothesis was that the median current health status at baseline/exposure 1 was exactly equivalent to the median current health status following exposure 3 to the intervention; p = 0.0332, Quantile Regression — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05; Random intercepts for subjects were included in the model; Median Difference (Net) = 13.10, 95% CI 2-sided [1.1 to 25.1] — This is the difference in median current health status between baseline/exposure 1 and exposure 3

9. Secondary Outcome: Number of Participants With Likely Low vs. Adequate Health Literacy According to SAHL-S&E Measurement
Description: Health literacy will be assessed using the short assessment of health literacy- Spanish. Scores range from 0 - 18 and a score above a 15 indicates that participants are likely to have adequate health literacy.
Time Frame: Baseline visit only
Population: 2 participants were withdrawn from the study by the PI and, therefore, their data are not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Participants
  Likely adequate health literacy | 16
  Likely low health literacy | 13
  Missing | 1

10. Secondary Outcome: Number of Participants With Likely Limited, Possibly Limited, or Adequate Health Literacy According to NVS Measurement
Description: A second measure of health literacy, the Newest Vital Sign (NVS) will also be administered. Scores on this scale range from 0-6 where a score of 0-1 suggests high likelihood of limited literacy, a score of 2-3 indicates the possibility of limited literacy, and a score of 4-6 almost always indicates adequate literacy.
Time Frame: Baseline visit only
Population: 2 participants were withdrawn from the study by the PI and, therefore, their data are not included in analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Participants
  Likely adequate health literacy | 5
  Possibility of limited health literacy | 11
  Likely limited health literacy | 14

11. Secondary Outcome: Number of Participants in Each Acculturation Category Presented in the Brief ARSMA
Description: The Brief Acculturation Rating Scale for Mexican Americans-II (Brief ARSMA)12 item instrument that assesses level of acculturation that has been used in Mexican Americans as well as other Latino subgroups, including Dominicans. Scores are calculated by summing the scores and dividing by 12 to get a mean acculturation. Higher scores indicate greater acculturation.
Time Frame: Baseline visit only
Population: 2 participants were withdrawn from the study by the PI and, therefore, were not included in analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Participants
  Very oriented to original culture | 13
  Oriented to original culture to approximately balanced bicultural | 6
  Slightly Anglo oriented bicultural | 4
  Strongly Anglo oriented | 4
  Very assimilated | 3

12. Secondary Outcome: Percent of Participants Who Complete an In-depth Qualitative Interview
Description: Participants will be invited to participate in an in-depth qualitative interview regarding their experiences. The number who participate will be reported as a percent of the total who are enrolled.
Time Frame: 6 months after baseline
Population: 2 participants were withdrawn from the study by the PI and, therefore, they are not included in analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Infographic Intervention Group
Number analyzed (Participants) | 30
Participants | 24

ADVERSE EVENTS:
Time Frame: Each participant was assessed while they were enrolled in the study, for up to 9 months (at 6-month visit) from baseline.
Description: We collected data for any adverse events that occurred during study-related activities.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
The global COVID-19 pandemic caused a research pause in mid-March 2020. This made it so that some of our participants were not able to complete their second out of three possible visits. Research activities were able to resume in May 2020 with strict COVID-19 safety measures in place. However, participants' third study visits were delayed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04102540/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04102540/ICF_002.pdf